CLINICAL TRIAL: NCT04780893
Title: A Randomized, Double Blind Sham Controlled, Pilot Study to Evaluate the Efficacy of Vestibular Nerve Stimulation (VeNS) for Sleep Management in People With Post- Traumatic Stress Disorder (PTSD).
Brief Title: Electrical Vestibular Nerve Stimulation (VeNS) as a Method of Sleep Management in People With PTSD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: New trial opportunity in the USA.
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: Clinical Trial Mentors (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: NIPTSD01
Record Dates: First submitted 2020-06-26; First posted 2021-03-04 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: PTSD; Sleep Disturbance; Insomnia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active VeNS (Active Comparator)
  Interventions: Device: Modius Sleep
- Sham VeNS (Sham Comparator)
  Interventions: Device: Modius Sleep

INTERVENTIONS:
Device: Modius Sleep — The device utilizes a technology called vestibular nerve stimulation (VeNS). The device will be placed on the head in a manner analogous to headphones and will deliver a small electrical current to the skin behind the ears, over the mastoid processes. Participants will be advised to use the device at home for 30 minutes per day.

SUMMARY:
This double blind randomized controlled study will enroll 20 subjects and will be conducted remotely. The study will be randomized for an 8-week period with a 1:1 active to sham device allocation. Primary endpoint analysis will be performed at 4 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Signed informed consent
2. Diagnosed PTSD by a medical practitioner
3. Post-Traumatic Checklist (PCL-5) score of 31 or above
4. Insomnia Severity Index (ISI) score of 15 or above
5. Male or female, age ≥ 18 years and ≤ 80 years at the time of signing informed consent
6. Ability and willingness to complete all study visits and procedures, including completion of mental health questionnaires
7. Ability and willingness to adhere to 30 minutes usage of the device daily for the duration of the study
8. No change to PTSD, mental health or insomnia medication within the past 3 months (regimen should be stable)
9. Agreement not to change usage of prescription or over the counter PTSD, mental health or insomnia medications for the duration of the study
10. Agreement not to undergo any significant lifestyle changes that may affect sleep (e.g., excessive exercise, sleep interventions etc.) for the duration of the study
11. Agreement not to use sleep trackers (e.g., Fitbit) for the duration of the study
12. Agreement not to travel across different time zones for the duration of the study
13. Access to Wi-Fi (to enable the study app to upload usage data)
14. Access to computer, laptop, iPad or tablet (to conduct remote study visits and complete study questionnaires remotely)
15. Willing to download and use Zoom (to conduct remote study visits)

Exclusion criteria:

1. History of skin breakdown, eczema, or other dermatological condition (e.g., psoriasis) affecting the skin behind the ears
2. Previous diagnosis of HIV infection or AIDS (HIV is known to cause vestibular neuropathy which would prevent VeNS from working)
3. Use of beta-blockers within 1 month of starting the study
4. A history of stroke or severe head injury as defined by a head injury that required a craniotomy or endotracheal intubation (in case this damaged the neurological pathways involved in vestibular stimulation)
5. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.)
6. Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using an adequate contraceptive method
7. Diagnosis of epilepsy
8. Diagnosis of active migraines
9. Previous use of Modius device
10. Participation in other research studies sponsored by Neurovalens
11. Participation in any other sleep or PTSD studies
12. Not fluent in English language
13. Have a member of the same household who is currently participating in this study
14. Failure to agree to use of device daily during study participation
15. History of vestibular dysfunction or other inner ear disease
16. Any other medical condition, or medication use, that in the opinion of the PI is likely to make the subject refractory to VeNS.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) score | 4 weeks
  To evaluate the effect of the Modius Sleep device, relative to control group on participants with insomnia. ISI is a self-report rating scale assessing the severity of insomnia symptoms (range 0-28) with higher scores indicating a more severe insomnia.

SECONDARY OUTCOMES:
PCL-5 Score | 4 weeks
  To evaluate the effect of the Modius Sleep device, relative to control group, on the symptoms of PTSD, quantified by change in the PCL-5 Score.
SF-36 Score | 4 weeks
  To evaluate the effect of the Modius Sleep device, relative to control group, on quality of life, quantified by change in the SF-36 Score.
Generalised Anxiety Disorder (GAD-7) Scores | 4 weeks
  To evaluate the effect of the Modius Sleep device, relative to control group, on anxiety, quantified by change in the GAD-7 score. GAD-7 is a self-report rating scale assessing the severity of anxiety (range 0-21), with higher score indicating more severe anxiety.
Prescription reduction | 4 weeks
  To evaluate the effect of the Modius Sleep device, relative to control group, on prescription reduction, quantified by change in medication.

CONTACTS AND LOCATIONS:
Overall Officials: David Wilson, MD, Principal Investigator — Clinical Trial Mentors

IPD SHARING:
Plan to Share IPD: No
Data will be transferred in an encrypted PDF format. Trial staff will be given direction on how to share the trial data and given access to one specific section of a controlled cloud service which is controlled via role based access. Once they have authenticated with the service and the service verifies that they have the correct role to access the system they will be directed to a single webpage within the application where they will be able to upload the encrypted PDF. This PDF is generated on the fly and is therefore not stored in another location that could become compromised. Generating the PDF on the fly means that the source data is extracted from the database, processed and delivered in the context of a single request. These data will be transferred for each subject when they complete participation in the study.